CLINICAL TRIAL: NCT00845026
Title: A Long-Term, Phase 2, Multicenter, Randomized, Open-Label Comparative Safety Study of LY2140023 Versus Atypical Antipsychotic Standard of Care in Patients With DSM-IV-TR Schizophrenia
Brief Title: A Safety Study Comparing LY2140023 to Atypical Antipsychotic Standard Treatment in Schizophrenic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12648; H8Y-MC-HBBR (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2022-09-01 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; pomaglumetad methionil; Aripiprazole; Olanzapine; Risperidone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2140023 (Experimental): LY2140023 (80 mg/day), given orally twice daily as two 40-mg tablets for 24 weeks
  Interventions: Drug: LY2140023
- aripiprazole (Active Comparator): aripiprazole (20 mg/day), given orally once daily for 24 weeks
  Interventions: Drug: aripiprazole
- olanzapine (Active Comparator): olanzapine (15 mg/day), given orally once daily for 24 weeks
  Interventions: Drug: olanzapine
- risperidone (Active Comparator): risperidone (4 mg/day), given orally, once or BID for 24 weeks
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: LY2140023 — 80 milligram (mg), oral tablets, twice daily: 40 mg in the morning, 40 mg in the evening, for 24 weeks. The dose may be adjusted to a minimum of 40 mg or a maximum of 160 mg.
  Other Names: pomaglumetad methionil
  Arms: LY2140023
Drug: aripiprazole — 10 mg, oral tablets, once a day in the evening for three days. Followed by a dose increase to 20 mg, 2-10 mg oral tablets, once a day in the evening, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 10 mg or a maximum of 30 mg (3-10 mg oral tablets).
  Other Names: Abilify
  Arms: aripiprazole
Drug: olanzapine — 10 mg dose (2-5 mg oral tablets) once every evening, for 3 days. Followed by an increase to 15 mg (3-5 mg oral tablets) once every evening, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 10 mg or a maximum of 20 mg (4-5 mg oral tablets).
  Other Names: Zyprexa
  Arms: olanzapine
Drug: risperidone — 2 mg dose, 2-1 mg oral tablets, given once or twice a day for 3 days. Followed by an increase to 4 mg (4-1 mg tablets), given once or twice a day, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 2 mg/day or a maximum of 6 mg/day (6-1 mg tablets).
  Other Names: Risperdal
  Arms: risperidone

SUMMARY:
The primary objective of this study was to assess time to discontinuation due to lack of tolerability among patients with schizophrenia receiving LY2140023, given orally twice daily for 24 weeks, versus those on atypical antipsychotic standard-of-care (SOC) treatment. Lack of tolerability was defined as discontinuation due to adverse events (AEs).

Patients who completed the active treatment phase were eligible to continue to an optional 28 weeks of treatment extension phase. This extension phase assessed key safety and efficacy measures.

DETAILED DESCRIPTION:
A Phase 2, multicenter, randomized, parallel, open-label study comparing the long-term safety and tolerability of LY2140023 with atypical antipsychotic agents considered to be the current SOC for patients with schizophrenia. The study included a 24-week active treatment phase and an optional 28-week active treatment extension phase.

The time to discontinuation due to AEs during Study Period III (24-week active treatment phase) was compared between LY2140023 and standard of care using the log-rank test from the Kaplan-Meier survival analysis. Patients who completed Study Period III or who discontinued for a reason other than AEs were considered as censored observations.

Secondary objectives were assessed during both Study Period III [Active Treatment Phase] and Study Period IV [Active Treatment Extension Phase]) except for treatment-emergent adverse events (TEAEs), extrapyramidal symptoms (EPS), electroencephalograms (EEGs), electrocardiograms (ECGs) (analysis for Study Period III only) (indicated in "Time Frame" in "Results" section)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Patients, in the investigator's opinion, must require a switch to another antipsychotic medication as clinically indicated or initiation of an antipsychotic agent
* Patients must be willing and able to be hospitalized, or to remain hospitalized (if already hospitalized), for up to 17 days
* The investigator expects, at the time of enrollment, that the patient will be able to be discharged from the hospital after the first 2 weeks of active treatment
* Disease symptoms must meet a certain range as assessed by the clinician
* Patients must have evidence of functional impairment (i.e. social or vocational deficiency)
* Patients must be considered reliable, have a level of understanding sufficient to perform all tests and examinations required by the protocol, and be willing to perform all study procedures
* Patients must be able to understand the nature of the study and have given their informed consent

Exclusion Criteria:

* Patients who are actively suicidal
* Patients who are pregnant or nursing
* Patients who have had electroconvulsive therapy (ECT) within 3 months of screening or who will have ECT at any time during the study
* Patients with uncorrected narrow-angle glaucoma, seizures, uncontrolled diabetes, certain diseases of the liver, uncontrolled thyroid condition or other serious or unstable illnesses
* Patients with Parkinson's disease, psychosis related to dementia or related disorders
* Patients with known Human Immunodeficiency Virus positive (HIV+) status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (23):
- United States (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willingboro, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amityville, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeSoto, Texas
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wiesbaden
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Russia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Khot'kovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lipetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nizhny Novgorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Samara

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included an antipsychotic drug taper/discontinuation (Study Period I) and a 3-day, single-blind placebo lead in (Study Period II). Study Period III was a 24-week active treatment phase. Participants who completed Study Period III were eligible to continue in an optional, 28-week, active treatment extension phase (Study Period IV).
Groups:
- Standard-of-Care (SOC): aripiprazole: 10 mg, oral tablets, once a day in the evening for three days. Followed by a dose increase to 20 mg, 2-10 mg oral tablets, once a day in the evening, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 10mg or a maximum of 30 mg (3-10 mg oral tablets).
  olanzapine: 10 mg dose (2-5 mg oral tablets) once every evening, for 3 days. Followed by an increase to 15 mg (3-5 mg oral tablets) once every evening, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 10 mg or a maximum of 20 mg (4-5 mg oral tablets).
  risperidone: 2 mg dose, 2-1 mg oral tablets, given once or twice a day for 3 days. Followed by an increase to 4 mg (4-1 mg tablets), given once or twice a day, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 2 mg/day or a maximum of 6 mg/day (6-1 mg tablets).
Period: Study Period III
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Started | 130 | 131
Completed | 35 (7 completed, left study; 28 completed, entered Study Phase IV.) | 59 (9 completed, left study; 50 completed, entered Study Phase IV.)
Not Completed | 95 | 72
Not completed — Adverse Event | 23 | 19
Not completed — Perceived lack of efficacy | 27 | 15
Not completed — Withdrawal by Subject | 19 | 15
Not completed — Entry Criteria not met | 8 | 11
Not completed — Lost to Follow-up | 4 | 5
Not completed — Protocol Violation | 8 | 1
Not completed — Scheduled conflict | 3 | 1
Not completed — Subject is moving or has moved | 2 | 4
Not completed — Transportation issues | 1 | 1
Period: Study Period IV
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Started | 28 (7 completed period III but left study; 28 completed period III AND entered period IV.) | 50 (9 completed period III, left study; 50 completed period III AND entered period IV.)
Completed | 12 | 46
Not Completed | 16 | 4
Not completed — Adverse Event | 4 | 0
Not completed — Perceived lack of efficacy | 2 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Entry Criteria Not Met | 1 | 0
Not completed — Subject is moving or has moved | 0 | 1
Not completed — Scheduling conflict | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- LY2140023: 80 mg, oral tablets, twice daily: 40 mg in the morning, 40 mg in the evening, for 24 weeks. The dose may be adjusted to a minimum of 40 mg or a maximum of 160 mg.
- Standard-of-Care (SOC): aripiprazole: 10 mg, oral tablets, once a day in the evening for three days. Followed by a dose increase to 20 mg, 2-10 mg oral tablets, once a day in the evening, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 10 mg or a maximum of 30 mg (3-10 mg oral tablets).
  olanzapine: 10 mg dose (2-5 mg oral tablets) once every evening, for 3 days. Followed by an increase to 15 mg (3-5 mg oral tablets) once every evening, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 10 mg or a maximum of 20 mg (4-5 mg oral tablets).
  risperidone: 2 mg dose, 2-1 mg oral tablets, given once or twice a day for 3 days. Followed by an increase to 4 mg (4-1 mg tablets), given once or twice a day, for 23 weeks and 4 days. The dose may be adjusted to a minimum of 2 mg/day or a maximum of 6 mg/day (6-1 mg tablets).
- Total: Total of all reporting groups
Arm/Group | LY2140023 | Standard-of-Care (SOC) | Total
Number analyzed (Participants) | 130 | 131 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.65 (10.87) | 39.45 (12.5) | 39.05 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 85 | 87 | 172
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 20 | 18 | 38
  Black or African American | 44 | 39 | 83
  Multiple | 1 | 3 | 4
  White | 65 | 71 | 136
Region of Enrollment [Number; unit: participants]
  United States | 58 | 59 | 117
  Mexico | 25 | 23 | 48
  Russian Federation | 41 | 45 | 86
  Germany | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Discontinuation Due to Adverse Event (AE)
Time Frame: Baseline through 24 weeks
Population: All randomized participants.
Measure: Mean (Standard Error); unit: days
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 130 | 131
days | 93.02 (5.95) | 116.86 (5.73)
Statistical Analysis 1: Comparison: LY2140023 vs Standard-of-Care (SOC); Test type: Superiority or Other; p = 0.184, Log Rank — No adjustments were made for multiplicity. All treatment comparisons were evaluated based on a two-sided significance level of 0.05

2. Secondary Outcome: Number of Participants With Shift From Baseline to Maximum Post-Baseline Grading in Electroencephalograms (EEGs)
Description: EEG scoring by a central neurologist is done by the following definitions: E0=Normal; E1(within normal)=fewer than 3 focal abnormalities or non-epileptiform abnormalities; E2(questionably epileptiform)=3-10 focal discharges and/or 1-10 multifocal or generalized discharges; E3=(clearly epileptiform)= Sharp/slow complex, runs of epileptiform abnormalities, greater than 10 total epileptiform discharges; and E4= seizure. Decreased= maximum (max) post-baseline (PB) EEG grading< baseline EEG grading; Increased= max PB EEG grading> baseline EEG grading; Same=no change from baseline to max PB result.
Time Frame: Baseline through 52 weeks
Population: All randomized participants with both baseline and at least one post-baseline value.
Measure: Number; unit: participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 103 | 118
participants
  Decreased | 11 | 8
  Same | 74 | 77
  Increased | 18 | 33

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in QT Intervals Electrocardiograms (ECGs)
Description: A potentially clinically significant QT interval (high) is defined as a value meeting the criteria of (> 450 millisecond [ms]) at anytime during the active treatment phase, provided it does not meet the criteria at baseline.
  (analysis for Study Period III only)
Time Frame: Baseline through 24 weeks
Population: All randomized participants with normal baseline measurement and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 118 | 127
participants | 3 | 4

4. Secondary Outcome: Number of Participants With Treatment-Emergent Change in Neurological Examination
Description: An increase in score from baseline was considered a treatment-emergent change, unless stated otherwise. Tremor: 0 (absent) - 3 (interferes with motor function); Nystagmus: 0 (absent) - 3 (present on forward gaze); Reflexes: 0 (absent) - 4 (clonic) with normal being a score 2, decrease or increase in score was considered change. Finger-nose and gait tests: 0 (normal) - 1(abnormal); Romberg's sign: (0) absent - (1) present; Muscular strength: 0 (no contraction)-5 (full/normal resistance), decrease in score was considered change; Myoclonic jerks: 0 (absent) - 3 (frequent).
Time Frame: Baseline through 52 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 130 | 131
participants
  Tremor | 16 | 23
  Nystagmus | 17 | 12
  Increased reflexes | 9 | 6
  Decreased reflexes | 20 | 28
  Abnormal finger-nose test | 2 | 0
  Romberg's sign | 0 | 1
  Abnormal Gait | 4 | 1
  Decreased muscle strength | 7 | 11
  Myoclonus | 1 | 0

5. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at 52 Weeks Endpoint
Description: Least Square (LS) Mean of change from baseline in BP is from a mixed model repeated measures (MMRM) model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline value and baseline-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 122 | 131
millimeters of mercury (mmHg)
  Supine Diastolic BP | 2.49 (2.09) | 0.87 (1.19)
  Standing Diastolic BP | 5.57 (2.06) | 1.10 (1.21)
  Supine Systolic BP | 2.84 (2.61) | 3.47 (1.63)
  Standing Systolic BP | 4.65 (2.65) | 1.93 (1.56)

6. Secondary Outcome: Change From Baseline in Weight at 52 Weeks Endpoint
Description: LS Mean of change from baseline in weight is from a MMRM model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline weight and baseline-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 122 | 131
kilogram (kg) | -4.76 (1.54) | 3.88 (1.08)

7. Secondary Outcome: Change From Baseline in Pulse Rate at 52 Weeks Endpoint
Description: LS Mean of change from baseline in pulse rate is from a MMRM model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline value and baseline-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 122 | 131
beats per minute (bpm)
  Supine Pulse | -1.62 (2.10) | -2.44 (1.22)
  Standing Pulse | -2.16 (2.16) | -2.41 (1.30)

8. Secondary Outcome: Number of Participants With Potentially Clinical Significant Change in Fasting Glucose Level
Description: Treatment-emergent changes in lab results on fasting glucose were analyzed using the American Diabetes Association (ADA 2001) and National Cholesterol Education Program (NCEP ATP III) guidelines. Glucose Normal to High is <100 milligram/deciliter (mg/dL) at baseline and ≥126mg/dL post-baseline.
Time Frame: Baseline through 52 weeks
Population: All randomized participants with a normal baseline and at least one post-baseline result.
Measure: Number; unit: participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 71 | 78
participants | 8 | 13

9. Secondary Outcome: Number of Participants With Potentially Clinical Significant Change in Lipids Level
Description: Treatment-emergent changes in lab results on lipids level were analyzed using the American Diabetes Association (ADA 2001) and National Cholesterol Education Program (NCEP ATP III) guidelines. Total cholesterol Normal to High is <200 mg/dL at baseline and ≥240 mg/dL post-baseline. Low-density lipoprotein (LDL) cholesterol Normal to High is <100 mg/dL at baseline and ≥160 mg/dL post-baseline. High-density lipoprotein (HDL) cholesterol Normal to Low is ≥40 mg/dL at baseline and <40 mg/dL post-baseline. Triglycerides Normal to High is <150 mg/dL at baseline and ≥200 mg/dL post-baseline.
Time Frame: Baseline through 52 weeks
Population: All randomized participants with a normal baseline and at least one post-baseline value.
Measure: Number; unit: participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 130 | 131
participants
  Total cholesterol Normal to High (n=56, 59): number analyzed (Participants) | 56 | 59
  Total cholesterol Normal to High (n=56, 59) | 3 | 6
  LDL cholesterol Normal to High (n=20, 22): number analyzed (Participants) | 20 | 22
  LDL cholesterol Normal to High (n=20, 22) | 0 | 0
  HDL cholesterol Normal to Low (n=74, 91): number analyzed (Participants) | 74 | 91
  HDL cholesterol Normal to Low (n=74, 91) | 16 | 23
  Triglycerides Normal to High (n=58, 77): number analyzed (Participants) | 58 | 77
  Triglycerides Normal to High (n=58, 77) | 7 | 21

10. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations Baseline Through 52 Weeks
Description: Columbia Suicide Rating Scale (C-SSRS): scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of participants with suicidal behaviors and ideations are provided. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation. There are no scores on a scale reported, rather, number of patients who reported "yes" as described above.
Time Frame: Baseline through 52 weeks
Population: All randomized participants with at least one post-baseline C-SSRS value.
Measure: Number; unit: participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 122 | 131
participants
  Suicidal ideation | 8 | 16
  Suicidal behavior/acts | 0 | 2

11. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at 52 Weeks Endpoint
Description: Assesses the positive and negative symptoms and general psychopathology associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210. LS Mean of change from baseline is from a mixed model repeated measures (MMRM) model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline score and baseline-by-visit interaction. Higher PANSS scores mean worse symptoms.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 119 | 128
units on a scale | -4.54 (4.22) | -21.47 (2.51)

12. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity Scale (CGI-S) at 52 Weeks Endpoint
Description: The CGI-S scale measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). LS Mean of change from baseline is from a MMRM model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline score and baseline-by-visit interaction. Higher CGI-S score means worse symptoms.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 121 | 131
units on a scale | -0.27 (0.25) | -0.81 (0.14)

13. Secondary Outcome: Change From Baseline in 16-Item Negative Symptoms Assessment (NSA-16) Total Score at 52 Weeks Endpoint
Description: The NSA-16 is used to rate behaviors (not psychopathology) associated with negative symptoms of schizophrenia and rates patients on 16 "anchors", each of which is rated 1 to 6. The total score is their sum and ranges from 16 to 96. Higher scores indicate greater severity of illness. LS Mean of change from baseline is from a MMRM model which includes treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline score and baseline-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 117 | 127
units on a scale | -2.86 (2.49) | -7.81 (1.58)

14. Secondary Outcome: Change From Baseline in Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery (MCCB): Overall Composite T-Score at 52 Weeks Endpoint
Description: The MCCB assesses cognitive function in 7 domains important in schizophrenia. The MCCB overall composite score is calculated by summing age- and gender-corrected T-scores of all the domains and then standardizing the sum to a T-score, where the mean is 50 and a standard deviation is 10. A higher score indicates better performance. LS Mean of change from baseline is from a MMRM model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline score and baseline-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 78 | 95
units on a scale | 5.29 (1.89) | 8.19 (1.27)

15. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at 52 Weeks Endpoint
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). LS Mean of changes from baseline is from a MMRM model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline score and baseline-by-visit interaction. Higher MADRS scores mean worse symptoms.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 117 | 128
units on a scale | 2.72 (1.40) | -2.82 (0.88)

16. Secondary Outcome: Change From Baseline in University of California-San Diego (UCSD) Performance-Based Skills Assessment-B (UPSA-B) Total Score at 52 Weeks Endpoint
Description: The UPSA-B is a performance-based assessment of improvement in functional capacity. Patients are asked to role-play tasks in 2 areas of functioning: communication and finances. Scores are assigned for each of the 2 subscales and a provided formulae is used to calculated an UPSA-B Total Score (range = 0-100). The higher score indicates a better performance. LS mean of change from baseline is from a MMRM model which includes the effects of treatment, gender, investigator site, visit, treatment-by-visit interaction, baseline score and baseline score by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 88 | 106
units on a scale | 11.82 (2.88) | 12.84 (1.69)

17. Secondary Outcome: Percentage of Participants With Response (Rate of Response) at 6 and 24 Weeks Endpoints
Description: Response is defined as reduction ≥ 30% from baseline on PANSS Total Score (Each PANSS item transformed to a 0-6 scale first). PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on an original scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210. Higher scores indicate greater severity of illness. (Analysis for Study Period III only)
Time Frame: 6 and 24 weeks
Population: All randomized participants with both baseline and at least one post-baseline PANSS values.
Measure: Number; unit: percentage of participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 120 | 128
percentage of participants
  6 weeks | 35.0 | 31.3
  24 weeks | 26.7 | 37.5

18. Secondary Outcome: Percentage of Participants With Remission (Rate of Remission) at Week 24 Endpoint
Description: Remission is defined as endpoint score of mild or better (≤3) for each of the following PANSS items: delusions, conceptual disorganization, hallucinatory behavior, social withdrawal, blunted affect, lack of spontaneity and flow of conversation, mannerisms and posturing, and unusual thought content. PANSS assesses the positive and negative symptoms and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated from 1 (symptom not present) to 7 (extremely severe). The sum of the 30 items is the PANSS total score and ranges 30 - 210. (Analysis for Study Period III only)
Time Frame: 24 weeks
Population: All randomized participants with both baseline and at least one post-baseline PANSS values.
Measure: Number; unit: percentage of participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 120 | 128
percentage of participants | 15.0 | 22.7

19. Secondary Outcome: Percentage of Participants With Relapse (Rate of Relapse)
Description: Relapse is defined as an increase in at least one PANSS positive item to a score>5 and an absolute increase of ≥2 points on that item post randomization , or hospitalization for any psychiatric condition, or active suicidal ideation or suicidal behavior as captured by the C-SSRS. PANSS assesses the positive and negative symptoms and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30-210.
Time Frame: Baseline through 52 weeks
Population: All randomized participants with non-missing relapse flag.
Measure: Number; unit: percentage of participants
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 130 | 131
percentage of participants | 26.2 | 16.8

20. Secondary Outcome: Change From Baseline in Subjective Well-Being Under Neuroleptic Treatment-Short Form (SWN-S) Total Score at 52 Weeks Endpoint
Description: Measures subjective well-being for previous 7 days. 20 items covering 5 health domains (subscales) (4 items each): emotional regulation, self-control, mental functioning, social integration, and physical functioning. Individual scores range from 1 (not at all) to 6 (very much). Subscale scores range from 4 to 24. Total score ranges from 20 to 120. LS mean of change from baseline is from a MMRM model which includes the effects of treatment, gender, investigator site, visit, treatment-by-visit interaction, baseline score and baseline score by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 106 | 120
units on a scale | 1.11 (2.83) | 4.15 (1.80)

21. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) at 52 Weeks Endpoint
Description: The Personal and Social Performance (PSP) scale is a 100-point, single-item, clinician-rated scale to assess 4 domains of functioning, including personal and social relationships, socially useful activities, self care, and disturbing and aggressive behaviors. Score ranges from 1-100. The higher score indicates a better health state. LS Mean of changes from baseline is from a MMRM model which includes the effects of treatment, gender, investigator site, visit, treatment-by-visit interaction, baseline score and baseline score by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 117 | 129
units on a scale | 6.47 (3.13) | 10.71 (1.89)

22. Secondary Outcome: Change From Baseline in EuroQoL Questionnaire-5 Dimension (EQ-5D) at 52 Weeks Endpoint
Description: The EQ-5D is a quality-of-life (QoL) instrument with 2 parts: a health status profile and a visual analog scale (VAS). The profile rates patients' health state in 5 domains and each of them ranges 1-3. The outcomes on the 5 domains are mapped to an index with range 0-1. The higher score indicates a better health state. The VAS is used to indicate the patient's health status with range 0=worst and 100=best. LS means are from a MMRM model with the effects of treatment, gender, investigator site, visit, treatment-by-visit interaction, baseline score and baseline score by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 130 | 131
units on a scale
  Visual Analog Scale (n=107, 120): number analyzed (Participants) | 107 | 120
  Visual Analog Scale (n=107, 120) | 4.83 (4.10) | 12.84 (2.43)
  Index Score (n=107, 119): number analyzed (Participants) | 107 | 119
  Index Score (n=107, 119) | 0.03 (0.05) | 0.10 (0.03)

23. Secondary Outcome: Change From Baseline in Number of Psychiatric Visits at 24 Weeks Endpoint
Description: Change in number of psychiatric visits between the 6 months prior to the active treatment phase and psychiatric visits reported during the active treatment phase was summarized. Treatment groups were compared on change using the analysis of covariance (ANCOVA) model. The model has baseline as a covariate, and investigative site, gender, and treatment as fixed effects. (Analysis for Study Period III only)
Time Frame: Baseline, 24 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: visits
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 103 | 112
visits | -2.60 (0.28) | -2.95 (0.27)

24. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Global Score at 52 Weeks Endpoint
Description: The BAS rates drug induced akathisia symptoms. Akathisia is rated on a 4-point scale, with 0 being no akathisia and 3 being severe akathisia. A global clinical assessment of akathisia is then scored on a 6-point scale, with 0 being no evidence of akathisia and 5 being severe akathisia. LS mean of change from baseline in BAS global score is from a MMRM model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline and baseline-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 122 | 131
units on a scale | -0.06 (0.05) | -0.08 (0.03)

25. Secondary Outcome: Change From Baseline in Simpson-Angus Scale (SAS) Total Score at 52 Weeks Endpoint
Description: The SAS is used to measure Parkinsonian type symptoms in patients exposed to antipsychotics. The scale consists of 10 items each rated on a 5-point scale, with 0 meaning complete absence of the condition and 4 meaning the presence of the condition in extreme form. The range of possible total score is 0-40. LS Mean of change from baseline in the SAS total score is from a MMRM model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline and baseline-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 121 | 131
units on a scale | -0.87 (0.26) | -0.82 (0.16)

26. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score at 52 Weeks Endpoint
Description: The AIMS is a 12-item scale designed to record the occurrence of dyskinetic movements. Items 1 to 10 are rated 0 - 4, with 0 being no dyskinetic movements and 4 being severe dyskinetic movements. Items 11 and 12 are yes/no questions regarding the dental condition of a subject. The total score is the sum of items 1-7 and ranges from 0-28. LS means of change from baseline in the AIMS total score is from a MMRM model which includes the effects of treatment, gender, investigative site, visit, treatment-by-visit interaction, baseline and baseline-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with both baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 | Standard-of-Care (SOC)
Number analyzed (Participants) | 122 | 131
units on a scale | 0.13 (0.29) | -0.23 (0.18)

ADVERSE EVENTS:
Time Frame: 1 year
Description: according to clinicaltrials.gov
Arm/Group | LY2140023 | Olanzapine | Aripiprazole | Risperidone
Serious Adverse Events (participants affected / at risk) | 22/130 | 6/48 | 4/48 | 2/35
Other Adverse Events (participants affected / at risk) | 96/130 | 32/48 | 40/48 | 28/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2140023 (N=130) | Olanzapine (N=48) | Aripiprazole (N=48) | Risperidone (N=35)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Psychotic behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 9 (9) | 3 (3) | 4 (4) | 1 (1)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2140023 (N=130) | Olanzapine (N=48) | Aripiprazole (N=48) | Risperidone (N=35)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (14) | 1 (1) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (19) | 2 (2) | 1 (1) | 2 (2)
Fatigue (General disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (10) | 1 (1) | 2 (2) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 12 (14) | 5 (6) | 7 (9) | 5 (7)
Blood triglycerides increased (Investigations) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 6 (6) | 1 (1) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (5) | 0 (0)
Akathisia (Nervous system disorders) | 2 (2) | 2 (2) | 5 (5) | 3 (3)
Extrapyramidal disorder (Nervous system disorders) | 3 (5) | 1 (1) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 17 (23) | 7 (8) | 2 (2) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Tremor (Nervous system disorders) | 5 (7) | 5 (8) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 10 (12) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 21 (28) | 5 (6) | 5 (8) | 4 (4)
Insomnia (Psychiatric disorders) | 21 (23) | 3 (3) | 6 (8) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 4 (5) | 3 (3) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 1/45 (1) | 1/13 (2) | 0/21 (0) | 1/10 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 2 (2) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days